CLINICAL TRIAL: NCT03007485
Title: A Comprehensive Disease Management Program to Improve Quality of Life in Disparity Hispanic and African-American Patients Admitted With Exacerbation of Chronic Pulmonary Diseases
Brief Title: Telehealth Pulmonary Rehabilitation for Hispanic and African-American Patients Admitted With Exacerbation of COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Negin Hajizadeh, Associate Professor of Medicine, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: AD-1511-33066
Record Dates: First submitted 2016-12-21; First posted 2017-01-02 (Estimated); Results first posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2021-12

CONDITIONS: COPD Exacerbation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Standard pulmonary rehabilitation
- Intervention (Experimental): Telehealth delivered pulmonary rehabilitation
  Interventions: Other: Telehealth Pulmonary Rehabilitation

INTERVENTIONS:
Other: Telehealth Pulmonary Rehabilitation — Exercise bikes equipped with software that enables a respiratory therapist to remotely conduct a pulmonary rehabilitation session with a patient while he or she is at home (or at a local community center). The patient's vital signs are continually monitored and the RT is able to remotely alert 911 if a patient is in distress. Educational videos and stretching exercises are also incorporated into this session to mimic what a standard pulmonary rehabilitation session offers.
  Arms: Intervention

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD), also known as emphysema, is the leading cause of hospitalization for older adults in the U.S., and a leading cause of death. Although there is no cure for COPD, a program called pulmonary rehabilitation (PR), which combines exercise and education, can help decrease re-hospitalizations and improve patients' quality of life. Unfortunately, very few COPD Latino and African-American patients actually get PR. These patients are unlikely to get referrals or to be able to attend PR due to lack of insurance, lack of transportation, or lack of a PR center in their area. Telehealth is a way of using computers to deliver healthcare long-distance, eliminating the need for a patient to travel to receive care. By using telehealth for PR, the patient can exercise on a stationary bike in his or her home, while being supervised by videoconference by a respiratory therapist (RT). The RT can "see" the patient, and deliver education by videoconference, and the patient can "see" the RT, so the patient does not need to leave home to get PR.

DETAILED DESCRIPTION:
Telehealth-delivered PR has been shown to be as effective as standard PR (patients go to an outpatient setting) at improving quality of life, and patients' exercise capacity. However, this has not been studied in the Latino and African-American population and it is not known how effective telehealth PR will be among this population.

For this study, the investigators hope to see if they can help COPD Latino and African-American patients with access to this needed resource through telehealth PR. They will compare standard PR and telehealth PR to determine if telehealth results in better outcomes for patients with moderate to severe COPD who were recently discharged from the hospital for COPD. The primary outcome the investigators will assess will be change in re-hospitalization rates. The secondary outcomes will include: change in quality of life, preparation to make decisions about clinical care, improved functional capacity, decreased dyspnea, anxiety, and depression.

The study will involve randomly assigning participants to make sure that they are just as likely to be in one group as the other to receive either: 1) referral for telehealth-delivered PR, or 2) referral to standard (outpatient) PR. Both PR programs consist of exercise and education twice a week for 8 weeks. The investigators will give the patients surveys to complete before they start the program and at the end of the program, to see if PR had any effect on the outcomes that are being measured. Patients will also be asked to participate in a qualitative interview and focus group to learn about the barriers they encountered even after receiving a referral to PR. These qualitative interviews will be conducted among a sample of participants representing those who withdrew, were lost-to-follow-up, completed PR and decided to only complete the surveys (i.e. not participate in PR).The investigators will enroll about 276 patients - with 138 patients in each group (telehealth PR or standard PR), so they can compare outcomes to see if telehealth PR was more, less, or equally effective as standard PR.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a diagnosis of COPD (defined by one pulmonary function tests (PFT) and who have not done pulmonary rehabilitation within the past 1 year and
* Hispanic or African-American (as defined by the patient him/herself).

Exclusion Criteria:

* individuals who completed PR in the past year or
* those unable to exercise or follow directions as determined by their outpatient pulmonologist/cardiologist or
* A diagnosis of dementia listed in the patient's electronic medical record
* Patients who weigh more than 300 pounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Negin Hajizadeh, MD, MPH, Principal Investigator — Hofstra Northwell School of Medicine, Northwell Health
Locations (1):
- Northwell Health, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poot CC, Meijer E, Kruis AL, Smidt N, Chavannes NH, Honkoop PJ. Integrated disease management interventions for patients with chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2021 Sep 8;9(9):CD009437. doi: 10.1002/14651858.CD009437.pub3. PMID 34495549
- [Derived] Pekmezaris R, Kozikowski A, Pascarelli B, Wolf-Klein G, Boye-Codjoe E, Jacome S, Madera D, Tsang D, Guerrero B, Medina R, Polo J, Williams M, Hajizadeh N. A Telehealth-Delivered Pulmonary Rehabilitation Intervention in Underserved Hispanic and African American Patients With Chronic Obstructive Pulmonary Disease: A Community-Based Participatory Research Approach. JMIR Form Res. 2020 Jan 31;4(1):e13197. doi: 10.2196/13197. PMID 32012039

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total 266 participants signed the informed consent and were randomized (131 to the TelePR arm and 135 to the SPR arm). Of the 131 randomized to TelePR, 20 were subsequently excluded after randomization because they no longer met inclusion criteria. Of the 135 randomized to SPR, 37 were excluded after randomization because they also no longer met inclusion criteria. Therefore, in total 209 participants were randomized and were included in the intention to treat analysis.
Groups:
- Telehealth-delivered Pulmonary Rehabilitation: Telehealth delivered pulmonary rehabilitation- Intervention
  Telehealth Pulmonary Rehabilitation: Exercise bikes equipped with software that enables a respiratory therapist to remotely conduct a pulmonary rehabilitation session with a patient while he or she is at home (or at a local community center). The patient's vital signs are continually monitored and the RT is able to remotely alert 911 if a patient is in distress. Educational videos and stretching exercises are also incorporated into this session to mimic what a standard pulmonary rehabilitation session offers.
Period: Overall Study
Arm/Group | Standard of Care | Telehealth-delivered Pulmonary Rehabilitation
Started | 98 | 111
Completed | 28 | 57
Not Completed | 70 | 54

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Intervention | Total
Number analyzed (Participants) | 98 | 111 | 209
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 48 | 91
  >=65 years | 55 | 63 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.96 (10.68) | 66.89 (10.80) | 66.42 (10.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 67 | 124
  Male | 41 | 44 | 85
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 41 | 48 | 89
  African-American | 57 | 63 | 120
Region of Enrollment [Number; unit: participants]
  United States | 98 | 111 | 209

OUTCOME MEASURES:

1. Primary Outcome: Composite of COPD Hospital Readmission/Death Within 6 Month of Discharge
Description: The investigators will analyze the change in the rate of patients' rehospitalizations following completion of pulmonary rehabilitation (PR). COPD Hospital Readmission were measured for Intention to Treat (ITT), medically cleared, and those who sat on the bike at least once. Composite of COPD hospital readmission or death within 6 months of discharge using all available (complete) data, and no imputation of missing data. Without adherence added, offset term omitted in the logistic regression.
Time Frame: 6 months post-discharge from hospitalization following COPD exacerbation
Population: TelePR and SPR arms were combined as pre-specified in the study protocol and explained below:
  The primary outcome was a composite of COPD-related hospital readmissions or death within 6 months of discharge. Logistic regression was used to compare the primary outcome in terms of the OR of event rates between arms, in 2 sets of models:
  * 1: Treatment arm only with no other covariates added to the model
  * 2: Treatment arm, adjusted for race and clinical site (stratification variables)
Measure: Number (95% Confidence Interval); unit: Hospitalizations/death
Groups:
- Intention to Treat (ITT): ITT: Total number of participants: 209 TelePR: 111 participants SPR: 98 participants
- Medically Cleared: Participants that were medically cleared by their pulmonologist and cardiologist (if needed) to participate in pulmonary rehab.
- Bike: Participants that agreed to participate, received medical clearance, and sat on the bike at least once.
Arm/Group | Intention to Treat (ITT) | Medically Cleared | Bike
Number analyzed (Participants) | 209 | 138 | 85
Hospitalizations/death
  Unadjusted | 1.34 [0.69 to 2.59] | 1.06 [0.43 to 2.58] | 0.88 [0.29 to 2.68]
  Adjusted (race, hospital) | 1.35 [0.69 to 2.66] | 1.09 [0.43 to 2.73] | 0.86 [0.27 to 2.72]
Statistical Analysis 1: Comparison: Intention to Treat (ITT) vs Medically Cleared vs Bike; Sample size and power calculation was a composite of COPD-related hospital readmissions or death within 6 months of discharge. First level of analysis was the ITT, which included all the patients randomly assigned to an arm at the beginning of the study (excluding those who were found to not meet inclusion criteria for referral). The second included all the patients medically cleared and third included all the patients who were medically cleared and who had participated in at least 1 PR session; Test type: Superiority; p < .05, t-test, 2 sided — Reported p-value was calculated; Odds Ratio (OR) = 1.0; The primary outcome was a composite of COPD-related hospital readmissions or death within 6 months of discharge (binary: yes/no). Logistic regression was used to compare the primary outcome in terms of the OR of event rates between the 2 arms, in 3 sets of models (per each of the 3 aforementioned level of analyses): * Model 1: Treatment arm only with no other covariates added to the model * Model 2: Treatment arm, adjusted for race and clinical site (stratification variables) * Model 3: Treatment arm, adjusted for race, clinical site, and risk factors reported in the literature to be associated with the primary outcome, for explanatory purposes To examine the role of adherence on the primary outcome, we included adherence as a binary variable and as a continuous variable (percentage of sessions attended) in the 3 models

2. Secondary Outcome: Functional Capacity Before and After Pulmonary Rehabilitation 6-minute Walk Test (SPR) Tested in Meters) Between Day 1 and 8-weeks
Description: The investigators will analyze the change in patients' functional capacity, as measured prior to beginning PR (Day 1), immediately following completion of PR (8 weeks). This measures the length the study participant walked/step (i.e. 2-minute step test (2MST)= how many steps the participant took, 6-minute walk test (6MWT)= the length the participant walked for in meters). Due to the limited space in TelePR participants home, they were only able to complete the 2MST, while SPR participants completed the 6MWT because the center had more space.
Time Frame: Prior to beginning PR (Day 1) and after completion of PR ( 8-weeks)
Population: Data in SPR arm reported in Outcome Measures in meters due to space.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Standard of Care
Number analyzed (Participants) | 37
Meters
  Day 1 | 261.92 (125.85)
  8 weeks | 275.29 (137.85)

3. Secondary Outcome: Change in Self-reported Quality of Life: Longitudinal Outcomes. Surveys Administered Over the Entire Follow up Period Directly Before and After the PR Program
Description: The investigators will analyze the change in patients' quality of life based on self-reported outcome measurements, as measured prior to beginning PR (Day 1), immediately following completion of PR (8 weeks), 6 months post-hospital discharge, 12 months post-hospital discharge.
  COPD Assessment Test (CAT): Maximal Score: 40, Minimal Score: 0; lower score denotes improvement
  Modified Medical Research Council Scale (MMRC): Maximal Score: 4, Minimal Score: 0; lower score denotes improvement
  All PROMIS scales have a maximal score of 20 and minimal score for all scales is 4; lower score denotes improvement.
Time Frame: Prior to beginning PR, after completion of PR, and 6 months and12 months post-discharge from hospitalizations following COPD exacerbation
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Telehealth-delivered Pulmonary Rehabilitation: Telehealth delivered pulmonary rehabilitation
  Telehealth Pulmonary Rehabilitation: Exercise bikes equipped with software that enables a respiratory therapist to remotely conduct a pulmonary rehabilitation session with a patient while he or she is at home (or at a local community center). The patient's vital signs are continually monitored and the RT is able to remotely alert 911 if a patient is in distress. Educational videos and stretching exercises are also incorporated into this session to mimic what a standard pulmonary rehabilitation session offers.
Arm/Group | Standard of Care | Telehealth-delivered Pulmonary Rehabilitation
Number analyzed (Participants) | 37 | 62
score on a scale
  COPD Assessment Test (CAT) Day 1 | 20.89 (8.53) | 22.37 (8.35)
  CAT 8-weeks | 20.18 (8.41) | 19.91 (7.94)
  CAT 6 months | 23.07 (7.54) | 21.12 (9.55)
  CAT 12 months | 20.09 (7.70) | 23.00 (8.26)
  Modified Medical Research Council Scale (MMRC) Day 1 | 2.24 (1.04) | 2.46 (1.16)
  MMRC 8-weeks | 2.24 (1.28) | 2.28 (1.14)
  MMRC 6 months | 2.48 (1.18) | 2.15 (1.30)
  MMRC 12 months | 2.45 (0.91) | 2.42 (1.20)
  PROMIS: Depression Day 1 | 7.38 (4.24) | 8.35 (4.21)
  PROMIS: Depression 8-weeks | 7.85 (3.78) | 7.97 (4.48)
  PROMIS: Depression 6 months | 9.25 (4.20) | 8.60 (4.28)
  PROMIS: Depression 12 months | 8.47 (4.25) | 8.29 (4.32)
  PROMIS: Fatigue | 9.70 (4.47) | 11.77 (4.95)
  PROMIS: Fatigue 8-weeks | 10.88 (4.21) | 10.43 (4.53)
  PROMIS: Fatigue 6 months | 11.43 (3.99) | 11.38 (4.90)
  PROMIS: Fatigue 12 months | 11.50 (4.68) | 10.92 (4.54)

4. Secondary Outcome: Functional Capacity Before and After Pulmonary Rehabilitation (2-minute Step Test (TelePR) Tested in Steps
Description: as for outcome 2
Time Frame: Prior to beginning PR (Day 1) and after completion of PR ( 8-weeks)
Population: Data in TelePR arm reported in Outcome Measures in steps due to space limitation.
Measure: Mean (Standard Deviation); unit: Steps
Groups:
- Telehealth-delivered Pulmonary Rehabilitation: Telehealth-delivered Pulmonary Rehabilitation
Arm/Group | Telehealth-delivered Pulmonary Rehabilitation
Number analyzed (Participants) | 62
Steps
  Day 1 | 43.87 (17.42)
  8 weeks | 51.12 (23.46)

5. Other Pre Specified Outcome: Measure of Patients' Uptake of PR i.e., Number of Referred Patients Who Participated in at Least One PR Session
Description: Given the improved convenience and access to PR, the investigators are looking to measure the degree to which patients adhere to their pulmonologists' referrals for pulmonary rehabilitation.
Time Frame: 8 weeks post-discharge from hospitalization following COPD exacerbation
Population: The denominator here is all patients who received a referral to PR.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Intervention
Number analyzed (Participants) | 98 | 111
Participants | 37 | 62

ADVERSE EVENTS:
Time Frame: Adverse Events was collected during the duration of the PR program - Day 1 to 8-weeks (completion of PR). The duration of time over which both, All-cause mortality and serious and other (non-serious) adverse events were assessed during Day 1 to 8 weeks (during PR) and until 6 months after enrollment into PR.
Description: Hospital readmission/death were monitored/assess within 6 month of discharged which includes the duration of PR 8 weeks. Adverse events were only collected during the duration of the PR program (Day1 to 8 weeks). Deaths were not assessed for a different duration of time than Serious and Other adverse events.
Arm/Group | Standard of Care | Telehealth-delivered Pulmonary Rehabilitation
All-Cause Mortality (participants affected / at risk) | 2/98 | 3/111
Serious Adverse Events (participants affected / at risk) | 3/98 | 3/111
Other Adverse Events (participants affected / at risk) | 3/98 | 13/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=98) | Telehealth-delivered Pulmonary Rehabilitation (N=111)
Serious Adverse Event (Cardiac disorders) | 1 | 3
Serious Adverse Event (Respiratory, thoracic and mediastinal disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=98) | Telehealth-delivered Pulmonary Rehabilitation (N=111)
Other (Not Including Serious) Adverse Events (Cardiac disorders) | 2 | 9
Other (Not Including Serious) Adverse Events (Eye disorders) | 1 | 1
Other (Not Including Serious) Adervse Events (Musculoskeletal and connective tissue disorders) | 0 | 2
Other (Not Including Serious) Adverse Events (Metabolism and nutrition disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-09): https://cdn.clinicaltrials.gov/large-docs/85/NCT03007485/Prot_SAP_000.pdf